CLINICAL TRIAL: NCT03681145
Title: Youth to Text or Telehealth for Engagement in HIV Care
Acronym: Y2TEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: California HIV/AIDS Research Program (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HD51-SF-060; T32DA007250 (NIH)
Record Dates: First submitted 2018-07-10; First posted 2018-09-21 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: HIV/AIDS; Mental Health Issue (E.G., Depression, Psychosis, Personality Disorder, Substance Abuse); Depression; Substance Use
Keywords: Young Adults; Telehealth; Health Disparity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression; Psychotic Disorders; Personality Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A-Intervention (Experimental): Participants will receive the study intervention immediately after study enrollment has been completed. The intervention will be delivered in 12, 20-30 minute sessions and text messaging over 4 months (1st session in person, remaining 11 sessions will be remote). The investigators will asses feasibility, acceptability and preliminary clinical outcomes of the Y2TEC intervention at 4 months and 6 months. During the waiting period, participants will receive text messages.
  Interventions: Behavioral: Counselor delivered telehealth intervention
- Group B-Wait-list (Experimental): Participants will be placed in a waitlist group for four months after study enrollment. Participants will receive the revised study intervention in 12, 20-30 minute sessions and text messaging over 4 months( all sessions remote). The investigators will asses feasibility, acceptability and preliminary clinical outcomes of the Y2TEC intervention at 4 months and 6 months. During the waiting period, participants will receive text messages.
  Interventions: Behavioral: Counselor delivered telehealth intervention

INTERVENTIONS:
Behavioral: Counselor delivered telehealth intervention — This is a technology-based counseling intervention for youth living with HIV (YLWH) focused on engagement in HIV care, mental health, and substance use challenges through text messaging and teleconferencing (telehealth). The intervention is delivered in 12 brief sessions.
  Other Names: Y2TEC

SUMMARY:
Youth To Text or Telehealth for Engagement in HIV Care (Y2TEC) is a randomized control pilot to assess the feasibility and acceptability of delivering a targeted problem-solving intervention to youth ages 18-29 living with HIV (YLWH) for improving HIV care engagement, mental health, and decreasing substance use. The intervention will be delivered to participants in two condition groups in remote telehealth sessions delivered via video-conference over 4 months. Participation in the study will last about 8 months.

The investigators hypothesize that the Y2TEC intervention will be feasible and acceptable for YLWH, and will result in improved HIV clinical outcomes. If feasible and acceptable, it can be scaled up for a multi-site randomized clinical trial and ultimately offered in the clinical care of YLWH.

DETAILED DESCRIPTION:
Due to a 50% increase in HIV-related deaths in youth from 2005 to 2012, there is a critical need for research to address health disparities in youth ages 18 to 29 years old living with HIV (YLWH) and for the tailoring of healthcare delivery to their unique and complex health needs. YLWH experience worse clinical outcomes than adults including high rates of mental health and substance use challenges that impact their medical care and adherence. Many YLWH have sub-optimal engagement in HIV care, including missed HIV provider visits and routine lab work. The consequence of suboptimal adherence in YLWH is increased risk of HIV transmission and a future generation of immunodeficient adults with drug-resistant virus. In response to this critical public health dilemma, the researchers propose to develop a telehealth intervention for YLWH focused on addressing engagement in HIV care, mental health, and substance use challenges. Telehealth holds promise in overcoming barriers to clinic attendance or research participation, such as transportation difficulties or HIV-related stigma concerns. Text messaging has also been used successfully for Antiretroviral therapy (ART) adherence and virologic suppression in African settings and has been examined in youth. The investigators have chosen these technology-based methods due to the presence of data supporting their efficacy, feasibility and acceptability, promise for future dissemination, limited research in YLWH, and ability to tailor based on patients' unique health needs. While these technologies can act on specific barriers to engagement in HIV care, they are inversely related in cost, burden to patient and provider, and intensity. Existing interventions for YLWH have been adapted to create the Youth to Text or Telehealth for Engagement in HIV Care Intervention (Y2TEC) through text messaging and teleconferencing (telehealth).

The Y2TEC telehealth intervention uses problem-solving therapy, a strengths-based orientation, and motivational interviewing to help participants identify and resolve potential barriers to engagement in HIV care and other barriers to overall wellness. Consisting of twelve 20-30 minute sessions with a trained social worker using a menu of structured sessions. Each session will focus on a specific topic as it relates to healthcare engagement and wellness, such as substance use, family support, or social support. The curriculum is designed increase engagement in HIV care and reduce viral loads. To achieve these outcomes, the behaviors most commonly targeted through the problem-solving activities will be related to medication adherence, attending clinic visits, and completing labs.

At the end of the study, the investigators will explore feasibility and acceptability using quantitative and qualitative methods. Participants will complete quantitative surveys at baseline, 4 months, 8 months, and study completion, as well as qualitative exit interviews conducted over the phone. Participants will consent to the study in person and will be randomized into one of two condition groups to receive the following: Group A: participants will immediately receive 1 brief counseling intervention in-person and 11 subsequent weekly sessions delivered remotely via video-conference and weekly text messaging. Then cross over to a waiting period receiving text messages for 12 weeks. Group B: Participants in the wait-list after consent and receive text messaging only for a period of 12 weeks then will receive a revised version of the intervention for 12 weeks with all sessions completed remotely via video-conference and text message.

The aims of this study are:

1. Employ: (1) mixed methods research to assess engagement in HIV care, technology use, substance use, and challenges with current systems of care among YLWH (18-29 years), (2) qualitative research to examine the perceptions of clinicians/managers of clinics and organizations serving YLWH on available referral services, system-wide barriers to care or referrals to substance use treatment, and age-specific challenges to patient care.
2. Develop a technology-based intervention for improving mental health and reducing substance for delivery in YLWH based on prior data and information learned in Aim 1.
3. Examine feasibility, acceptability, and preliminary clinical outcomes of the technology-based intervention among YLWH on improved engagement in HIV care and mental health, and reduced substance use.

The investigators hypothesize that the Y2TEC intervention will be feasible and acceptable for YLWH. Our secondary hypotheses: H1: Antiretroviral adherence, engagement in care, and CD4+ cell count will be higher and HIV RNA levels will be lower in the intervention arm (Group A) relative to the wait-list arm (Group B) at 4 months. H2: Among those enrolling in the study with a detectable HIV RNA, there will be a minimum of 1log10 reduction in HIV RNA at 4 months among the intervention arm and at 8 months among the wait-list arm relative to baseline and 4 months, respectively. H3: Among those enrolling in the study with an undetectable HIV RNA, there will be a maintenance of virologic suppression at 4 months among the intervention arm and at 8 months among the wait-list control arm relative to baseline and 4 months, respectively.

The investigators postulate parallel hypotheses for self-reported ART adherence, appointment attendance based on medical records, and self-reported composite of engagement in care with mean levels of these variables being highest in the Telehealth arm and lowest in the control arm. Conversely, the screener for substance use (CRAFFT score) should be highest in the control arm and lowest in the Telehealth arm. If this innovative intervention is found to be feasible and acceptable, it can be scaled up for a multi-site adaptive randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* HIV+
* Youth (18-29 years)
* Living or receiving health care in the eastern region of the San Francisco Bay Area (i.e.

East Bay)

* Willing and able to provide informed consent
* Access to a mobile phone with text messaging capability
* Access to the internet through a mobile phone, computer or tablet

Exclusion Criteria:

The Investigators will exclude those with evidence of severe cognitive impairment or active psychosis that may impede the ability to provide informed consent.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Feasibility: Participant Retention at 4 months | 4 months
  Percentage of participants retained in the study at 4 months
Feasibility: Mean Number of Teleconference Disconnections | 8 months
  Mean of one disconnection per videoconferencing session
Feasibility: Video Quality | 4 months
  1 item, Likert scale (0-10) (0= poor quality; 10= excellent quality) To calculate feasibility by video quality, the investigators will report the average score among all users.
Feasibility: Sound Quality | 4 months
  1 item, Likert scale (0-10) (0= poor quality; 10= excellent quality) To calculate feasibility by sound quality, the investigators will report the average score among all users.
Feasibility: Participant Response Time to Text | 8 months
  Mean number of days between bi-directional text message and participants' response
Acceptability: Measure participant satisfaction of the telehealth intervention as assessed by use of original 30-item satisfaction survey | 8 months
  Measure participant satisfaction with the telehealth intervention at 8-months using a 30-item questionnaire (1 Excellent-6 Unsatisfied) administered through an online survey. An average score greater than or equal to 144 (80%) will be considered acceptable.
Acceptability: Measure participant satisfaction of the telehealth sessions from 0 to 8 months via 2-item scale adapted from Session Rating Scale (SRS) | 8 months
  Measure participant satisfaction of each telehealth session via 2-item scale adapted from Session Rating Scale (SRS) (1-Strongly Agree to 4 Strongly Disagree, lower rating indicates higher satisfaction) administered by text-messaging. Average participant satisfaction over 12 telehealth sessions from baseline to 8 months.
Feasibility: Participant Retention at 8 months | 8 months
  Percentage of participants retained in the study at 8 months

SECONDARY OUTCOMES:
Clinical Impact: Self-reported medication adherence | 8 months
  Measure changes in participants' self-reported medication adherence based on 1-item adherence rating (1-Excellent- 6 Poor, lower rating indicates higher adherence) from baseline to 8 months.
Clinical Impact: Frequency of Substance Use | 0 to 8 months
  Measure participants' change in substance use from baseline to 8 months using a 10-item questionnaire adapted from the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) administered through an online survey to measure frequency of participants' substance use. Scoring range is 0-Never to 6 almost daily, lower rating indicates lower substance use.
Severity of Substance Use from 0 to 8 months | 0 to 8 months
  Measure participants' changes in substance use from baseline to 8 months using the Drug Abuse Screening Test (DAST), a 10-item questionnaire administered through an online survey to measure severity of participants' substance use. Responses are summed. Scoring (0-10);0-2 Low substance use, 9-10 Severe substance use.
Alcohol Use | 0 to 8 months
  Measure participants' alcohol use from baseline to 8 months using the Alcohol Use Disorder Test (AUDIT), a 10-item questionnaire administered through an online survey to measure severity of participants' alcohol use. Responses are summed. Scoring range is 0-20+; 0-7 Low alcohol use, 20+ High dependence.
Clinical Impact: Depression | 0 to 8 months
  Measure participants' depression from baseline to 8 months using the Patient Health Questionnaire ( PHQ-9), a 9-item Likert scale score (0 - 3) 0 "not at all", 3 "nearly every day". Responses are summed. Scores will have a range of 0-27. PHQ-9 scores of > 10 are associated with moderate to severe depression.
Clinical Impact: Post Traumatic Stress Disorder (PTSD) | 0 to 8 months
  Measure participants' self-reported PTSD from baseline to 8 months using the Psychopathy Checklist-revised (PCL), a 20-item Likert questionnaire administered through an online survey. Scoring: 0 points for "not at all", 1 point for "a little bit", 2 points for "moderately", 3 points for "quite a bit", 4 points for "extremely".Scores will have a range of 0-80. Responses are summed.
Measure participant HIV Knowledge using HIV Treatment Knowledge Scale | 0 to 8 months
  Assess participants' knowledge of HIV from baseline to 8 months through the HIV Treatment Knowledge measure, a 15-item self-report questionnaire. Scoring out of 15 (0-11 Inadequate, 12-15 Adequate). Scores will have a range of 0-15.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco Mission Hall, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wootton AR, Legnitto DA, Gruber VA, Dawson-Rose C, Neilands TB, Johnson MO, Saberi P. Telehealth and texting intervention to improve HIV care engagement, mental health and substance use outcomes in youth living with HIV: a pilot feasibility and acceptability study protocol. BMJ Open. 2019 Jul 16;9(7):e028522. doi: 10.1136/bmjopen-2018-028522. PMID 31315868
- [Result] Saberi P, Ming K, Dawson-Rose C. What does it mean to be youth-friendly? Results from qualitative interviews with health care providers and clinic staff serving youth and young adults living with HIV. Adolesc Health Med Ther. 2018 Apr 24;9:65-75. doi: 10.2147/AHMT.S158759. eCollection 2018. PMID 29731672
- [Result] Saberi P, Dawson Rose C, Wootton AR, Ming K, Legnitto D, Jeske M, Pollack LM, Johnson MO, Gruber VA, Neilands TB. Use of technology for delivery of mental health and substance use services to youth living with HIV: a mixed-methods perspective. AIDS Care. 2020 Aug;32(8):931-939. doi: 10.1080/09540121.2019.1622637. Epub 2019 May 28. PMID 31132864
- [Result] Saberi P, McCuistian C, Agnew E, Wootton AR, Legnitto Packard DA, Dawson-Rose C, Johnson MO, Gruber VA, Neilands TB. Video-Counseling Intervention to Address HIV Care Engagement, Mental Health, and Substance Use Challenges: A Pilot Randomized Clinical Trial for Youth and Young Adults Living with HIV. Telemed Rep. 2021 Jan 7;2(1):14-25. doi: 10.1089/tmr.2020.0014. eCollection 2021. PMID 33575683
- [Result] Wootton AR, McCuistian C, Legnitto Packard DA, Gruber VA, Saberi P. Overcoming Technological Challenges: Lessons Learned from a Telehealth Counseling Study. Telemed J E Health. 2020 Oct;26(10):1278-1283. doi: 10.1089/tmj.2019.0191. Epub 2019 Dec 3. PMID 31800368